CLINICAL TRIAL: NCT01370889
Title: Pilot Study of Resveratrol in Postmenopausal Women With High Body Mass Index
Brief Title: Resveratrol in Postmenopausal Women With High Body Mass Index
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: NCI-2011-02593; NCI-2011-02593 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000701405; 10-0653-04 (Other: University of Arizona Health Sciences Center); UAZ08-12-01 (Other: DCP); P30CA023074 (NIH); N01CN35158 (NIH); NCT02022332 (obsolete NCT alias)
Record Dates: First submitted 2011-06-09; First posted 2011-06-10 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-04

CONDITIONS: Healthy, no Evidence of Disease
MeSH Terms: interventions — Resveratrol

ARMS (1):
- Basic Science (resveratrol) (Experimental): Patients receive resveratrol PO QD for 12 weeks.
  Interventions: Drug: resveratrol; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: resveratrol — Given PO
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot phase I trial studies resveratrol in postmenopausal women with high body mass index. Chemoprevention is the use of certain drugs to keep cancer from forming. The use of resveratrol may keep cancer from forming. Studying samples of blood and urine in the laboratory from postmenopausal women who are taking resveratrol may help doctors learn more about the effects of resveratrol on biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the effect of pharmacological doses of resveratrol on serum estradiol levels in post-menopausal women with high body mass index (BMI).

SECONDARY OBJECTIVES:

I. Assess the effect of resveratrol on serum estrone, testosterone, and sex hormone-binding globulin (SHBP).

II. Assess the effect of resveratrol on serum levels of insulin and C-peptide. III. Assess the effect of resveratrol on adipocytokine expression and secretion as measured by serum leptin and adiponectin.

IV. Assess the effect of resveratrol on inflammatory cytokines as measured by serum C-reactive protein (CRP).

V. Assess the effect of resveratrol on oxidative stress as measured by urinary 8-isoprostaglandin F2 alpha (8-iso-PGF2 alpha) and 8-hydroxydeoxyguanosine (8OHdG).

VI. Assess the safety of resveratrol intervention as measured by reported adverse events, complete blood count with differential (CBC/diff), comprehensive metabolic panel (CMP), and lipid profile.

VII. Assess the relationship between systemic study agent exposure and biomarker modulation.

OUTLINE:

Patients receive resveratrol orally (PO) once daily (QD) for 12 weeks.

After completion of study therapy, patients are followed up for 2 weeks

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women with a body mass index (BMI) of 25 kg/m^2 or greater
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1; Karnofsky 70% or above
* Leukocytes >= 3,000/uL
* Absolute neutrophil count (ANC) >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 2.0 mg/dL
* Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) =< 1.5 times upper limit of normal (ULN)
* Creatinine =< 1.0 times ULN
* Ability and willingness to limit resveratrol-containing foods to no more than one serving each per day for about 14 weeks
* Negative mammogram or negative workup of mammographic findings within prior 12 months prior to enrollment for women >= 50 years of age
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Have had invasive cancer(s) within the past 5 years except non-melanoma skin cancer
* Within 3 months of or concurrent usage of any other investigational agents
* History of allergic reactions attributed to resveratrol
* Unwilling or unable to refrain from taking herbal medicines and dietary supplements
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Within 3 months of or concurrent estrogen or progesterone replacement therapy, oral contraceptives, androgens, luteinizing hormone-releasing hormone analogs, prolactin inhibitors, or antiandrogens; vaginal estrogen is acceptable.

Within 3 months of or concurrent usage of tamoxifen, raloxifene, other selective estrogen-receptor modulators, or aromatase inhibitors

* Regular usage (more than 2 times a week) of estrogenic supplements or herbal remedies (e.g., Remifemin, black cohosh, red clover, dong quai, soy isoflavones, dehydroepiandrosterone [DHEA], flaxseed, diindolylmethane [DIM], genistein, and daidzein) within the past 3 months or concurrently; dietary consumption of phytoestrogens/isoflavones (such as soy, tofu, millet, barley, natto, tempeh, miso, soy milk, soy sauce) is acceptable as these sources are not concentrated
* Concurrent use of anti-diabetic drugs such as:

  * Insulin
  * Sulfonylureas (e.g., glipizide, glyburide, or glimepiride)
  * Meglitinides (e.g., repaglinide or nateglinide)
  * Biguanides (e.g., metformin)
  * Thiazolidinediones (e.g., rosiglitazone or pioglitazone)
  * Alpha-glucosidase inhibitors (e.g., acarbose or miglitol)
  * Dipeptidyl peptidase-4 (DPP-4) inhibitors (e.g., sitagliptin)
* Concurrent use of warfarin or phenytoin

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Change in serum estradiol levels in postmenopausal women with high BMI | From baseline to 12 weeks (post-intervention)
  A two-sided paired t-test will be performed to determine whether the change is significant at a significance level of 5%. If the data distribution indicates non-normality or skewedness in violation of the assumptions of the t-test, non-parametric tests will be used. Linear regression techniques will be used to adjust for potential confounders, e.g. age and BMI.

SECONDARY OUTCOMES:
Change in serum estrone | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in serum testosterone | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in serum sex hormone-binding globulin (SHBG) | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in serum levels of insulin | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in serum levels of C-peptide | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in serum leptin | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in serum adiponectin | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in inflammatory markers, measured by serum C-reactive protein | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in urinary 8-iso-PGF2alpha | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Change in urinary 8OHdG | From baseline to 12 weeks (post-intervention)
  Similar statistical analysis procedures as described for the primary endpoint will be performed to evaluate the changes of each of the endpoints at a significance level of 5%. Analysis will not be corrected for multiple comparisons but results will be interpreted cautiously. If the data distribution indicates non-normality or skewness, non-parametric tests will be used.
Incidence of reported adverse events | Up to 12 weeks
  Descriptive statistics of the type and frequency of all adverse events will be generated, including 95% confidence intervals.
Incidence of changes in CBC/diff, blood chemistry, and lipids | Up to 12 weeks
Study agent/metabolite levels | Up to 12 weeks
  The Spearman correlation coefficient will be calculated to evaluate the correlation between biomarker changes and study agent/metabolite levels. Linear regression techniques will be used to adjust for potential confounders, e.g. age and BMI.

CONTACTS AND LOCATIONS:
Overall Officials: Hsiao-Hui (Sherry) Chow, Principal Investigator — University of Arizona Health Sciences Center
Locations (2):
- United States (2):
  - Arizona Cancer Center - Tucson, Tucson, Arizona
  - University of Arizona Health Sciences Center, Tucson, Arizona

REFERENCES:
- [Derived] Chow HH, Garland LL, Heckman-Stoddard BM, Hsu CH, Butler VD, Cordova CA, Chew WM, Cornelison TL. A pilot clinical study of resveratrol in postmenopausal women with high body mass index: effects on systemic sex steroid hormones. J Transl Med. 2014 Aug 14;12:223. doi: 10.1186/s12967-014-0223-0. PMID 25115686